CLINICAL TRIAL: NCT03156595
Title: Demonstrate the Value of Using Hypnosis in Chimiotherapy- Induced Chronic Neuropathies
Acronym: NHYP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRIP 2015 - HUS n°6395
Record Dates: First submitted 2017-03-09; First posted 2017-05-17 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Chemotherapy-induced Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse interview (Placebo Comparator): Personal interview with nurses to evaluate the relief of neuropathic pains with the reference treatment. (If necessary send to the medical team ) It's a listening time around neuropathic pain which altered the quality of life.
  Interventions: Behavioral: Nurse interview
- Hypnosis session (Experimental): Hypnosis sessions with nurses or psychologists, with deepening sessions to facilitate self-hypnosis learning.
  Interventions: Behavioral: Hypnosis sessions

INTERVENTIONS:
Behavioral: Nurse interview — Personal interview with nurses to evaluate the relief of neuropathic pains with the reference treatment. (If necessary send to the medical team ) It's a listening time around neuropathic pain which altered the quality of life.
  Other Names: Listening time
  Arms: Nurse interview
Behavioral: Hypnosis sessions — Hypnosis sessions with a nurse or psychologist, with deepening sessions to facilitate self-hypnosis learning.
  Arms: Hypnosis session

SUMMARY:
Chimiotherapy produces neuropathies injuries to 30% to 70% cases. A third of those patients keeps suffering from this side effects disabilities and their quality of life is seriously affected.

Hypnosis, as a non-invasive tool without physical side effects, might be used to relieve them.

the purpose of this trial based on our own experience, is to demonstrate the value of using hypnosis and self-hypnosis in chimiotherapy- induced chronic neuropathies.

The aim will be to sustainably improve the quality of life by expanding self-management of pain and motor function side effect.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age :18 years
* Chemiotherapy- induced chronic neuropathies for at least 2 months with a DN4 score >4
* Failure of classic treatment used to relief neuropathic
* Having stopped chemotherapy treatment and being in complete or partial response or in tumoral stability
* Without any planed chemiotherapy during the study
* Having signed a written informed consent.
* French efficient understanding
* With health insurance coverage
* availability during all the study
* With efficient contraception for women of childbearing age

Exclusion Criteria:

* No participation to another study at the same time
* Suffering from neuropathy before having chemotherapy
* Other disease that may cause neuropathy
* deafness
* Any medicine that could cause neuropathy
* Neurological or psychiatrical disease past or present
* Mental retardation
* Allergy to EMG's electrodes
* Unable to consent, under tutelage or curatorship or judiciary safeguard
* Pregnant or nursing woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2017-08-04 (Actual); Primary Completion 2021-11-04 (Estimated); Study Completion 2021-11-04 (Estimated)

PRIMARY OUTCOMES:
Measure at 12 weeks (D84) benefits of hypnosis and self-hypnosis on the sensitive dimension of the quality of life of patients with chronic peripheral neuropathies arising from a cancer chemotherapy and inadequately relief with reference treatments. | Day 84

SECONDARY OUTCOMES:
Measure at 12 weeks (D84) benefits of hypnosis and self-hypnosis on the motor dimension of the quality of life of patients with chronic peripheral neuropathies arising from a cancer chemotherapy and inadequately relief with reference treatments. | Day 84
Measure at 12 weeks (D84) benefits of hypnosis and self-hypnosis on the loss of autonomy of patients with chronic peripheral neuropathies arising from a cancer chemotherapy and inadequately relief with reference treatments. | Day 84
Measure benefits of hypnosis on the neuropathic pain intensity | Day 28, day 56 and Day 84.
Measure benefits of hypnosis on a psychotropic treatments | Day 0, Day 28, day 56 and Day 84.
Measure benefits of hypnosis on analgesic treatments | Day 0, Day 28, day 56 and Day 84.
Measure benefits of hypnosis on tendon reflexes, deep and superficial sensitivity, muscular strength | Day 84
Measure benefits of hypnosis on electrophysiological abnormalities related to neuropathy | Day 84
Measure benefits of hypnosis on self- hypnosis in the experimental group | Day 28, Day 56 and D84
Evaluate the safety in the two arms, due to hypnosis adverse effects, to pain treatment or another reason | Day 0, Day 28, Day 56, Day 84 and in case of serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Caroline MAURER, Nurse, Study Chair — Strasbourg's University Hospitals; Raoul HERBRECHT, MD, Principal Investigator — Strasbourg's University Hospitals
Locations (1):
- University Strasbourg Hospital, Strabsourg, France

IPD SHARING:
Plan to Share IPD: No